CLINICAL TRIAL: NCT01688583
Title: The Effectiveness and Tolerability of Fentanyl Matrix in Chronic Non-cancer Pain; Assessment of Patient's Pain Treatment Goal Achievement: Multicenter, Prospective, Open-label, Observational Study
Brief Title: The Effectiveness and Tolerability of Fentanyl Matrix in Chronic Non-cancer Pain; Assessment of Patient's Pain Treatment Goal Achievement
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100728; FENPAI4094 (Other: Janssen Korea, Ltd., Korea); FEN-KOR-5045 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Chronic non-cancer pain; Fentanyl matrix; Transdermal system
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Fentanyl matrix
  Interventions: Drug: Fentanyl matrix

INTERVENTIONS:
Drug: Fentanyl matrix — Dose will be adjusted in accordance with patient's degree of pain and treatment response in the investigator's judgment.

SUMMARY:
The purpose of this study is to assess the effectiveness and tolerability of Fentanyl matrix in chronic non-cancer pain.

DETAILED DESCRIPTION:
This is a multicenter, prospective (a study in which the patients are identified and then followed forward in time for the outcome of the study), open-label (all people know the identity of the intervention), observational study intended to examine the effectiveness of Fentanyl matrix through the degree of improvement of pain. Fentanyl matrix is a transdermal (through the skin) system providing continuous delivery of fentanyl for 72 hours. Fentanyl matrix will be administered to patients with chronic (prolonged) non-cancer pain under routine practice during 12 weeks. Dose will be adjusted in accordance with patient's degree of pain and treatment response in the investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

* Complain of chronic non-cancer pain that persists for >= 3 months
* Pain inadequately controlled by previous treatment with narcotic analgesics (opium or opium-like compounds with potent analgesic effects, eg, tramadol, codeine, morphine, oxycodone)
* Women must be postmenopausal, surgically sterile, abstinent, or practicing an effective method of birth control if they have childbearing potential
* Male patients who agree to use a method of birth control and not to donate sperm for 1 month after the last dose of the study drug
* A written informed consent for study participation

Exclusion Criteria:

* Experience of treatment with Fentanyl matrix within the past 4 weeks
* No previous experience of use of narcotic analgesics
* Past or current history of alcohol or drug abuse
* Cannot use transdermal analgesics due to skin disorder
* Have serious psychiatric disorder and cannot complete overall study procedures and questionnaire in the judgment of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who complain of chronic pain and have pain inadequately controlled by previous treatment with narcotic analgesics (eg, tramadols, codeines, morphines, oxycodone), and are judged to require Fentanyl matrix administration will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with mean % Pain Intensity Difference (%PID) >= 50% from baseline to endpoint | 12 weeks
  Pain intensity will be measured using a numeric rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
The change from baseline in mean pain intensity | Baseline, Week 12
  Pain intensity will be measured using a numeric rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
The difference between the patient's pain treatment goal set at baseline | Baseline, Week 12
  The degree of pain the patient wishes to achieve by the end of treatment, set at baseline. The degree of pain will be measured using a numeric rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
The degree of night sleep disturbance due to pain | 12 weeks
  Sleep disturbance due to pain will be measured using a Numeric Rating Scale (NRS): 1 = None, 10 = Complete.
The degree of Interference with Daily Life Performance due to Pain | 12 weeks
  The degree of interference with daily life performance due to pain will be assessed on a 5-point scale: 1 = No interference, 5 = Great interference. Daily life performance means household work performance, etc.
The degree of Interference with Social Life Performance due to Pain | 12 weeks
  The degree of interference with social life performance due to pain will be measured on a 5-point scale; 1 = No interference, 5 = Great interference. Social life performance means interpersonal relationship, going out, working life, etc.
The patient's global assessment of pain treatment | 12 weeks
  The patient will assess on a 5-point scale (1= not effective, 5= greatly effective) how effective the study drug has been in the judgment of the study participant.
The investigator's global assessment of pain treatment | 12 weeks
  The investigator will assess on a 5-point scale (1= not effective, 5= greatly effective) how effective the study drug has been for a patient, in the judgment of the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (11):
- South Korea (11):
  - Andong
  - Busan
  - Daegu
  - Daejeon
  - Goyang
  - Incheon
  - Jeonju
  - Kwangiu
  - Kwanju
  - Seoul
  - Wŏnju